CLINICAL TRIAL: NCT06153524
Title: The Effect of Increasing Physical Activity or Reducing Mobile Phone Use on Mental Health in Young People in Austria: a Randomised Controlled Trial
Brief Title: The Effect of Increasing Physical Activity or Reducing Mobile Phone Use on Mental Health in Young People in Austria
Acronym: SPARKY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danube University Krems (Other)
Collaborators: University of Innsbruck (Unknown); University of Vienna (Other)
Responsible Party: Principal Investigator, Rachel Dale, Dr, Danube University Krems
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3757
Record Dates: First submitted 2023-11-13; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Mental Health Issue
Keywords: intervention; adolescent; exercise; Fitbit; smartphone; depression; well-being
MeSH Terms: conditions — Motor Activity; Depression | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A three-arm randomised controlled trial
Masking Description: Due to the nature of the interventions, no blinding can be involved
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical Activity (Experimental): The PA group will be guided by sports scientists to progressively build up to 60-minutes of daily moderate-vigorous exercise. The goals will be tailored to existing activity levels so as not to increase physical activity too quickly and will be set out in an action plan to be handed out at the beginning of the intervention. For the autonomous PA plan, participants from the PA group will be given Fitbits and a comprehensive manual of instructions to help them build their own weekly plan, and they will participate in weekly online meetings. The manual is structured with four main sections: 1. General information on training, 2. Moderate activity, 3. Vigorous activity, 4. Training agenda. The latter is for the participants to fill in after every training session. This information is then cross-checked by the PA specialists with the comments gathered during the weekly meetings.
  Interventions: Behavioral: Physical activity
- Smartphone (Experimental): The ST group will be guided by psychologists/psychotherapists to reduce their average daily phone use by 50% over the first two months of the intervention and to maintain this for the final month, and this will be measured using a screen time recording application. This intervention group will receive a list of nudge strategies (adapted from Olson et al., 2022) to add small barriers which guide them into reducing their phone use (e.g. disabling notifications, not using phone in bed). Participants will select three strategies (minimum) to try in the first month, then an additional two (minimum) for the second month. They will also receive a list of potential replacement activities to do instead of using their phone and are asked to choose which activities they want to try and/or list their own ideas. How easy/difficult each strategy is, how enjoyable the replacement activities are, and whether they want to change will be discussed in the meetings.
  Interventions: Behavioral: Smartphone time
- Control (No Intervention): The control group will receive basic written explanatory information on the study and will then simply record all their physical activity and screen time, without being set specific goals. This group will receive a list of mental health resources, all materials for increasing physical activity and reducing screen time and will be invited to a psychoeducation talk at the end of the study.

INTERVENTIONS:
Behavioral: Physical activity — 12x weekly advice sessions and autonomous physical activity to gradually build up moderate-vigorous exercise.
  Arms: Physical Activity
Behavioral: Smartphone time — 12x weekly advice sessions and autonomous use of replacement activities and strategies to gradually reduce daily smartphone use.
  Arms: Smartphone

SUMMARY:
Introduction: Data show adolescent mental health has declined in recent years, possibly due to increased uncertainty and loss of opportunities. The SPARKY study aims to test an at-home intervention which aims to promote autonomous healthy levels of physical activity and smartphone use, in turn reducing clinical mental illness symptoms and increasing wellbeing.

Methods and analysis: Adolescents (14-19 years) in Austria and Germany will be recruited and randomised into one of three groups (physical activity, smartphone, control). The physical activity (PA) and smartphone time (ST) groups will be guided over 12-weeks to increase PA or decrease ST respectively. All groups will objectively measure PA using wrist-worn trackers and ST using an app and will regularly self-report on standardised mental health scales. Analyses will be run to assess the pre-post changes in mental health in the intervention groups compared to the control.

Ethics and dissemination: The conduct of the trial was approved by the institutional research ethics board and written informed consent will be obtained from participants and the parents of those under 18. Data will be stored open access. Findings will be disseminated through conferences, media interviews and publications to peer-reviewed journals.

Overall, mental health interventions are sorely needed in adolescents to counteract the effects of the pandemic and other uncertainties. The at-home nature of the intervention will promote autonomous healthy habit formation in youth.

DETAILED DESCRIPTION:
Design: A three-arm randomised controlled trial with a physical activity group, a smartphone-use group and a control group. Outcome assessments are to be conducted at baseline, biweekly during the intervention, at three months (post-intervention), and at one month, six months and one year post-intervention (follow-ups). The study is not blinded.

Hypotheses:

The predictions can be divided into two categories: 1. improvements in mental health and 2. assessing behaviour change. All hypotheses are directional.

1. Mental health:

   * The primary hypothesis is that the intervention groups will show a greater improvement in their mental health than the control group from pre- to post-intervention.
   * Secondly, it is predicted that these improvements in mental health will be sustained at the follow-up stage.
   * Thirdly, those individuals who meet the goals will have better mental health than those who do not.
2. Behaviour change:

   * As a measure of the success of the intervention, it is predicted that those in the intervention groups will be more likely to meet the physical activity and screen time goals at post-intervention and follow-up than the control group.
   * Finally, it can be predicted that merely tracking daily activity and screen time is enough to promote some behaviour change and therefore it is predicted that the control group will be more likely to meet the goals at post-intervention than pre-intervention.

ELIGIBILITY:
Inclusion Criteria:

* aged 14-19
* own a smartphone
* use their phones more than 4 hours per days
* do less than 60 minutes of vigorous sport on 3 days per week and/or less than 60 minutes of moderate activity on 5 days per week.
* conduct work/school in German
* hair at least 1cm long

Exclusion Criteria:

* should not be in current medical care or have physical constraints which affect movement.
* should not have a diagnosis of schizophrenia/psychotic disorder, substance use disorder, symptoms of an eating disorder (≥2 positive answers on SCOFF questionnaire).
* should not have dyed hair. Participants will complete an online screening questionnaire to assess eligibility for inclusion.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in depression score over time | pre-baseline, post-baseline (baseline = 2-weeks), every other week during the intervention period (12 weeks), at immediately at post-intervention (intervention = 12-weeks) and at 1-month, 6-months and 1-year post-intervention
  Depression will be assessed using the 9-item self-report Patient Health Questionnaire (PHQ-9, validated in German). Items refer to the last two weeks and are rated on a 4-point Likert scale from not at all (0) to nearly every day (3). The scores range from 0-27 and cut-offs of ≥11 for those 18 or under and ≥10 for those over 18 indicate clinically relevant symptoms.
  Measured in all three groups online via the ESMira app.
Change in anxiety score over time | pre-baseline, post-baseline (baseline = 2-weeks), every other week during the intervention period (12 weeks), at immediately at post-intervention (intervention = 12-weeks) and at 1-month, 6-months and 1-year post-intervention
  Anxiety will be measure using the self-report Generalized Anxiety Disorder Scale (GAD-7; validated in German). The seven items on a four-point scale can result in a maximum score of 21 and the cut-offs for clinically relevant symptoms are ≥11 in those 18 and under and ≥10 in over 18s. Measured in all three groups online via the ESMira app.
Change in well-being score over time | pre-baseline, post-baseline (baseline = 2-weeks), every other week during the intervention period (12 weeks), at immediately at post-intervention (intervention = 12-weeks) and at 1-month, 6-months and 1-year post-intervention
  Well-being will be assessed using the World Health Organisation-five well-being index (WHO-5; validated in German) which consists of five items with scores ranging from 0 (no well-being) to 100 (maximal well-being). Measured in all three groups online via the ESMira app.

SECONDARY OUTCOMES:
Change in happiness score over time | pre-baseline, post-baseline (baseline = 2-weeks), every other week during the intervention period (12 weeks), at immediately at post-intervention (intervention = 12-weeks) and at 1-month, 6-months and 1-year post-intervention
  Happiness will be assessed using the Cantril ladder whereby participants are asked to rate the status of their lives on a scale of 1 (hopeless) to 10 (prospering). Measured in all three groups online via the ESMira app.
Change in sleep quality over time | ISI-7 at pre-baseline and immediately at post-intervention (intervention=12weeks).
  Sleep quality will be assessed with the Insomnia Severity Index (ISI-7; validated in German), a 5-point scale with a score of ≥22 representing severe insomnia symptoms. ISI-7 measured in all three groups online via the ESMira app.
Change in sleep duration over time | daily during baseline period (2 weeks), daily during intervention period (12 weeks) and daily during 1-month, 6-month and 1-year follow-ups (1 week each)
  Sleep duration will be assessed using the Fitbit Inspire 3 devices. While Fitbits are not as accurate as polysomnography, recent-generation models perform fairly well at estimating sleep parameters and will therefore be used for within-subject pre-post assessments but not for inter-group comparisons. Sleep duration measured daily via Fitbit tracker.
Change in perceived stress score over time | pre-baseline, post-baseline (baseline = 2-weeks), every other week during the intervention period (12 weeks), at immediately at post-intervention (intervention = 12-weeks) and at 1-month, 6-months and 1-year post-intervention
  Stress will be assessed using the Perceived Stress Scale (PSS-10; validated in German); a 10-item questionnaire with five-point scales. PSS-10 measured in all groups online via the ESMira app.
Change in cortisol levels over time | pre-baseline & post-intervention (14 weeks: 2-week baseline + 12-week intervention)
  Hair cortisol as a biomarker for chronic stress will be assessed. Hair samples will be collected by the participants themselves and sent by post.
Change in smartphone addiction over time | pre-baseline, post-baseline (baseline = 2-weeks), every other week during the intervention period (12 weeks), at immediately at post-intervention (intervention = 12-weeks) and at 1-month, 6-months and 1-year post-intervention
  Participants will complete the Smartphone Addiction Scale - short version (SAS-SV; validated in German). This scale is 10 items scored from 1-6 resulting in a maximum score of 60. The cut-off score considered as a smartphone addiction in adolescents is 31 for boys and 33 for girls. SAS-SV measured in all groups online via the ESMira app.
Change in smartphone usage over time | measured daily via the ESMira app over baseline period (2 weeks), during the intervention period (12 weeks) and daily during 1-month, 6-month and 1-year follow-ups (1 week each)
  Time spent using the smartphone will be assessed with an objective app to measure daily overall screen time (ESMira).
Change in physical activity over time | Measured daily via Fitbit trackers over baseline period (2 weeks), during the intervention period (12 weeks) and daily during 1-month, 6-month and 1-year follow-ups (1 week each).
  Physical activity will primarily be measured using the Fitbit Inspire 3 devices. The Fitbit app designates activities as light, moderate or vigorous. Time spent in moderate and vigorous activity will be recorded. Furthermore, the question "on how many days in the last week were you physically active for at least 60 minutes" will be asked. This allows comparison to data previously collected on youth.
Qualitative measures | 1 x per week during the intervention period (12 weeks)
  Qualitative measures will include content analysis of the weekly online meetings, which will be recorded for this purpose. The discussions each week will be free but will include the same overall structure (see interventions section). The first and last sessions will include additional questions for qualitative analysis: e.g. what are your current burdens/stressors? What is your current mood?

OTHER OUTCOMES:
Intervention acceptability | Measured once immediately at post-intervention (intervention = 12 weeks)
  Intervention acceptability will be measured using the German ZUF-8 questionnaire. The eight items are on a four-point scale with sum scores ranging from 8-32, with a higher score representing higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Dale, PhD, Principal Investigator — University for Continuing Education Krems
Locations (1):
- University for Continuing Education Krems, Krems, Lower Austria, Austria

IPD SHARING:
Plan to Share IPD: Yes
Anonymised quantitative data will be stored open access on the DOOR repository of the University for Continuing Education Krems.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available upon publication of the accompanying manuscripts and will remain online.
Access Criteria: Open access
URL: https://www.donau-uni.ac.at/de/universitaet/service/bibliothek/publikationsservices/door.html

REFERENCES:
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] Lowe B, Kroenke K, Herzog W, Grafe K. Measuring depression outcome with a brief self-report instrument: sensitivity to change of the Patient Health Questionnaire (PHQ-9). J Affect Disord. 2004 Jul;81(1):61-6. doi: 10.1016/S0165-0327(03)00198-8. PMID 15183601
- [Background] Richardson LP, McCauley E, Grossman DC, McCarty CA, Richards J, Russo JE, Rockhill C, Katon W. Evaluation of the Patient Health Questionnaire-9 Item for detecting major depression among adolescents. Pediatrics. 2010 Dec;126(6):1117-23. doi: 10.1542/peds.2010-0852. Epub 2010 Nov 1. PMID 21041282
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Lowe B, Decker O, Muller S, Brahler E, Schellberg D, Herzog W, Herzberg PY. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. Med Care. 2008 Mar;46(3):266-74. doi: 10.1097/MLR.0b013e318160d093. PMID 18388841
- [Background] Klein EM, Brahler E, Dreier M, Reinecke L, Muller KW, Schmutzer G, Wolfling K, Beutel ME. The German version of the Perceived Stress Scale - psychometric characteristics in a representative German community sample. BMC Psychiatry. 2016 May 23;16:159. doi: 10.1186/s12888-016-0875-9. PMID 27216151
- [Background] Haghayegh S, Khoshnevis S, Smolensky MH, Diller KR, Castriotta RJ. Accuracy of Wristband Fitbit Models in Assessing Sleep: Systematic Review and Meta-Analysis. J Med Internet Res. 2019 Nov 28;21(11):e16273. doi: 10.2196/16273. PMID 31778122
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Kwon M, Kim DJ, Cho H, Yang S. The smartphone addiction scale: development and validation of a short version for adolescents. PLoS One. 2013 Dec 31;8(12):e83558. doi: 10.1371/journal.pone.0083558. eCollection 2013. PMID 24391787
- [Background] Schmidt J, Lamprecht F, Wittmann WW. [Satisfaction with inpatient management. Development of a questionnaire and initial validity studies]. Psychother Psychosom Med Psychol. 1989 Jul;39(7):248-55. German. PMID 2762479
- [Background] Dale R, Jesser A, Pieh C, O'Rourke T, Probst T, Humer E. Mental health burden of high school students, and suggestions for psychosocial support, 1.5 years into the COVID-19 pandemic in Austria. Eur Child Adolesc Psychiatry. 2023 Jun;32(6):1015-1024. doi: 10.1007/s00787-022-02032-4. Epub 2022 Jul 28. PMID 35900473
- See also: Pre-registration of the study plan following open science principles — https://osf.io/m5wzv